CLINICAL TRIAL: NCT01583426
Title: A Randomized Phase III Trial Comparing Nanoparticle-based Paclitaxel With Solvent-based Paclitaxel as Part of Neoadjuvant Chemotherapy for Patients With Early Breast Cancer (GeparSepto)
Brief Title: Nanoparticle-based Paclitaxel vs Solvent-based Paclitaxel as Part of Neoadjuvant Chemotherapy for Early Breast Cancer (GeparSepto)
Acronym: GeparSepto
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GBG Forschungs GmbH (Other)
Collaborators: Celgene Corporation (Industry); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GBG 69; 2011-004714-41 (EudraCT Number)
Record Dates: First submitted 2012-04-18; First posted 2012-04-24 (Estimated); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Tubular Breast Cancer Stage II; Mucinous Breast Cancer Stage II; Breast Cancer Female NOS; Invasive Ductal Breast Cancer; Tubular Breast Cancer Stage III; HER-2 Positive Breast Cancer; Inflammatory Breast Cancer Stage IV; Inflammatory Breast Cancer
Keywords: GeparSepto; GBG 69; GBG; German Breast Group; neo-adjuvant; GBG Forschungs GmbH; Tubular breast cancer stage II; Mucinous breast cancer stage II; Invasive ductal breast cancer; Tubular breast cancer stage III; HER-2 positive breast cancer; Inflammatory breast cancer
MeSH Terms: conditions — Carcinoma, Ductal, Breast; Inflammatory Breast Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- nab-Paclitaxel (Experimental): nab-Paclitaxel (125 mg/m² weekly, infusion) is applicated for 12 weeks, followed by epirubicin and cyclophosphamide, applicated 4 cycles 3-weekly . In case of HER2-positive tumor patients receive tarstuzumab and pertuzumab 3-weekly during all cycles.
  Interventions: Drug: nab-Paclitaxel
- Paclitaxel (Active Comparator): Paclitaxel (80 mg/m² weekly, infusion) is applicated for 12 weeks, followed by epirubicin and cyclophosphamide, applicated 4 cycles 3-weekly . In case of HER2-positive tumor patients receive tarstuzumab and pertuzumab 3-weekly during all cycles.
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: nab-Paclitaxel — nab-Paclitaxel 125 mg/m² weekly for 12 weeks
  Other Names: Abraxane
  Arms: nab-Paclitaxel
Drug: Paclitaxel — Paclitaxel 80 mg/m² weekly for 12 weeks
  Arms: Paclitaxel

SUMMARY:
Current guidelines as those from the AGO-Breast commission recommend for neoadjuvant breast cancer patients either a sequence of 4 cycles EC followed by 4 cycles of a taxane or 6 cycles of TAC based on previous large scale studies.

Treatment of patients with HER2-positive disease should include also simultaneous application of trastuzumab.

Solvent-based taxanes (paclitaxel, docetaxel) cause severe toxicities not only by the active agents itself but also by the solvents like cremophor. Nab-paclitaxel (Abraxane®) is a solvent-free formulation of paclitaxel encapsulated in albumin. It does not require premedication with corticosteroids or antihistamines to prevent the risk of solvent-mediated hypersensitivity reactions. This new formulation improves safety profile, allows higher dosing with shorter infusion duration, and produces higher tumor drug concentration.

As neoadjuvant treatment does not only allow to compare competing treatment approaches with a very high quality (homogenous treatment population, precise assessment of response by histological assessment), but also to identify predictive markers, this trial will compare weekly nab-paclitaxel with solvent-based paclitaxel at their currently optimal doses.

In case of HER2-positive tumor status patients receive Pertuzumab and Trastuzumab additionally.

DETAILED DESCRIPTION:
Primary Objectives:

To compare the pathological complete response (pCR=ypT0 ypN0) rates of neoadjuvant treatment of nab-paclitaxel with solvent-based paclitaxel as part of neoadjuvant treatment of operable or locally advanced primary breast cancer

Secondary Objectives:

* To assess the pCR rates per arm separately for the stratified subpopulations.
* To determine the rates of ypT0/is ypN0; ypT0 ypN0/+; ypT0/is ypN0/+; ypT(any) ypN0; and regression grades.
* To determine the response rates of the breast tumor and axillary nodes based on physical examination and imaging tests (sonography, mammography, or MRI) after treatment in both arms.
* To assess clinical response rate after taxane in both groups
* To determine the breast conservation rate after each treatment.
* To assess the toxicity and compliance.
* To assess the time of onset of grade 3 neuropathy
* To assess the time of resolution of grade 3/4 neuropathy to at least grade 1
* To determine loco-regional invasive recurrence free survival (LRRFS), distant-disease-free survival (DDFS), invasive disease-free survival (IDFS), and overall survival (OS) in both arms and according to stratified subpopulations.
* To assess regional recurrence free survival (RRFS) in patients with initial node-positive axilla converted to negative at surgery and treated with sentinel node biopsy alone.
* To determine the pCR rate and local recurrence free survival (LRFS) in patients with a clinical complete response (cCR) and a negative core biopsy before surgery.
* To examine and compare pre-specified molecular markers such as SPARC, gp60, calveoline 1 and other markers potentially differentially predicting efficacy of nab-paclitaxel and solvent-based paclitaxel on core biopsies before, during and after chemotherapy.

Objectives of Substudies:

* To assess, characterize, and correlate circulating tumor cells and proteins with the effect of treatment (CTC Substudy).
* To correlate Single Nucleotide Polymorphisms (SNPs) of genes with the associated toxicity and histologically assessed treatment effect (Pharmacogenetic substudy)
* To assess ovarian function measured by amenorrhea rate in correlation with changes in E2, FSH, LH , Anti-Müller Hormone, ultrasound-follicle count in patients aged < 45 years.

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible for study participation only if they comply with the following criteria:

* Written informed consent for all study according to local regulatory requirements prior to beginning specific protocol procedures.
* Complete baseline documentation must be sent to GBG Forschungs GmbH.
* Unilateral or bilateral primary carcinoma of the breast, confirmed histologically by core biopsy. Fine-needle aspiration alone is not sufficient. Incisional biopsy is not allowed. In case of bilateral cancer, the investigator has to decide prospectively which side will be evaluated for the primary endpoint.
* Tumor lesion in the breast with a palpable size of >= 2 cm or a sonographical size of >= 1 cm in maximum diameter. The lesion has to be measurable in two dimensions, preferably by sonography. In case of inflammatory disease, the extent of inflammation can be used as measurable lesion.
* Patients must be in the following stages of disease:

  * - cT2 - cT4a-d or
  * cT1c and cN+ or
  * - cT1c and pNSLN+ or
  * - cT1c and ER-neg and PR-neg or
  * - cT1c and Ki67 > 20%
  * - cT1c and HER2-pos
  * In patients with multifocal or multicentric breast cancer, the largest lesion should be measured.
* Centrally confirmed ER/PR/HER-2, Ki-67 and SPARC status detected on core biopsy. ER/PR positive is defined as >1% stained cells and HER2-positive is defined as IHC 3+ or in-situ hybridisation (ISH) ratio >2.0. Formalin-fixed, paraffin-embedded (FFPE) breast tissue from core biopsy has therefore to be sent to the Dept. of Pathology at the Charité, Berlin prior to randomization.
* Age >= 18 years.
* Karnofsky Performance status index >= 80%.
* Normal cardiac function must be confirmed by ECG and cardiac ultrasound (LVEF or shortening fraction) within 3 months prior to randomization. Results must be above the normal limit of the institution. For patients with HER2-positive tumors LVEF must be >= 55%.
* Laboratory requirements:
* Hematology
* - Absolute neutrophil count (ANC) >= 2.0 x 109 / L and

  * Platelets >= 100 x 109 / L and
  * Hemoglobin >= 10 g/dL (>= 6.2 mmol/L)
* Hepatic function
* - Total bilirubin < 1.5x UNL and

  * ASAT (SGOT) and ALAT (SGPT) <= 1.5x UNL and
  * Alkaline phosphatase <= 2.5x UNL.
* Negative pregnancy test (urine or serum) within 14 days prior to randomization for all women of childbearing potential.
* Complete staging work-up within 3 months prior to randomization. All patients must have bilateral mammography, breast ultrasound (<= 21 days), breast MRI (optional), chest X-ray (PA and lateral), abdominal ultrasound or CT scan or MRI, and bone scan done. In case of positive bone scan, bone X-ray is mandatory. Other tests may be performed as clinically indicated.
* Patients must be available and compliant for central diagnostics, treatment and follow-up.

Exclusion Criteria:

* Prior chemotherapy for any malignancy.
* Prior radiation therapy for breast cancer.
* Pregnant or lactating patients. Patients of childbearing potential must implement adequate non-hormonal contraceptive measures (barrier methods, intrauterine contraceptive devices, sterilization) during study treatment.
* Inadequate general condition (not fit for anthracycline-taxane-targeted agents-based chemotherapy).
* Previous malignant disease without being disease-free for less than 5 years (except CIS of the cervix and non-melanomatous skin cancer).
* Known or suspected congestive heart failure (>NYHA I) and / or coronary heart disease, angina pectoris requiring antianginal medication, previous history of myocardial infarction, evidence of transmural infarction on ECG, uncontrolled or poorly controlled arterial hypertension (i.e. BP >160 / 90 mm Hg under treatment with two antihypertensive drugs), rhythm abnormalities requiring permanent treatment, clinically significant valvular heart disease.
* History of significant neurological or psychiatric disorders including psychotic disorders, dementia or seizures that would prohibit the understanding and giving of informed consent.
* Persons who have been admitted to an institution by order of jurisdictional or governmental grounds.
* Pre-existing motor or sensory neuropathy of grade 2 or more by NCI-CTC criteria v 4.0.
* Currently active infection.
* Definite contraindications for the use of corticosteroids.
* Known hypersensitivity reaction to one of the compounds or incorporated substances used in this protocol.
* Concurrent treatment with:
* - chronic corticosteroids unless initiated > 6 months prior to study entry and at low dose (10 mg or less methylprednisolone or equivalent).
* - sex hormones. Prior treatment must be stopped before study entry.
* - other experimental drugs or any other anti-cancer therapy.
* Participation in another clinical trial with any investigational, not marketed drug within 30 days prior to study entry.
* Male patients.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1229 (Actual)
Dates: Start 2012-07; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Pathological complete response (pCR=ypT0 ypN0) rates of neoadjuvant treatment of nab-paclitaxel with solvent-based paclitaxel as part of neoadjuvant treatment of operable or locally advanced primary breast cancer. | 24 weeks (time window + 3 weeks)
  No microscopic evidence of residual invasive or non-invasive viable tumor cells in all resected specimens of the breast and axilla.
  Pathological response will be assessed considering all removed breast and lymphatic tissues from all surgeries.
  The primary endpoint will be summarized as pathological complete remission rate for each treatment group.

SECONDARY OUTCOMES:
Rates of ypT0/is ypN0; ypT0 ypN0/+; ypT0/is ypN0/+; ypT(any) ypN0, and regression grade | 24 weeks (time window + 3 weeks)
  Response (by physical examination, imaging response, breast conservation) will also be summarized as rates in each treatment group.
Clinical and imaging response | 24 weeks (time window + 3 weeks)
  To determine the response rates of the breast tumor and axillary nodes based on physical examination and imaging tests (sonography, mammography, or MRI) after treatment in both arms.
Tolerability and safety | during treatment (24 weeks)
  Descriptive statistics for the 4 treatments (each taxane +/- anti-HER2-treatment) will be given on the number of patients whose treatment had to be reduced, delayed or permanently stopped.
pCR rates per arm | 24 weeks (time window + 3 weeks)
  To assess clinical response rate after taxane in both groups.
Breast conservation rate | 24 weeks (time window + 3 weeks)
  To determine the breast conservation rate after each treatment.
Onset of grade 3 neuropathy | 24 weeks (time window + 3 weeks)
  To assess the time of onset of grade 3 neuropathy.
Resolution of grade 3/4 neuropathy | 24 weeks (time window + 3 weeks)
  To assess the time of resolution of grade 3/4 neuropathy to at least grade 1.
Regional recurrence free survival (RRFS) in patients with initial node-positive axilla | until event occurs - no event for cured patients
  To assess regional recurrence free survival (RRFS) in patients with initial node-positive axilla converted to negative at surgery and treated with sentinel node biopsy alone.
pCR rate and local recurrence free survival (LRFS) in patients with a clinical complete response (cCR) and a negative core biopsy | 24 weeks (time frame + 3 weeks)
  To determine the pCR rate and local recurrence free survival (LRFS) in patients with a clinical complete response (cCR) and a negative core biopsy before surgery.
Examination and comparison of molecular markers | Baseline, 12 weeks and 24 weeks (time frame + 3 weeks)
  To examine and compare pre-specified molecular markers such as SPARC, gp60, calveoline 1 and other markers potentially differentially predicting efficacy of nab-paclitaxel and solvent-based paclitaxel on core biopsies before, during and after chemotherapy.
  The aim is to identify potential predictive short and long term parameters.
CTC Substudy | Baseline, 12 weeks and 24 weeks (time frame + 3 weeks)
  To assess, characterize, and correlate circulating tumor cells and proteins with the effect of treatment.
Pharmacogenetic substudy | Baseline
  To correlate Single Nucleotide Polymorphisms (SNPs) of genes with the associated toxicity and histologically assessed treatment effect.
Ovarian substudy | Baseline, 6 months, 12 months, 18 months, 24 months 30 months
  To assess ovarian function measured by amenorrhea rate in correlation with changes in E2, FSH, LH , Anti-Müller Hormone, ultrasound-follicle count in patients aged <45 years.
Loco-regional invasive recurrence free survival (LRRFS) in both arms and according to stratified subpopulations. | 5 years
  LRRFS is defined as the time period between registration and first event and will be analyzed after the end of the study by referring to data from GBG patient's registry.
Distant-disease-free survival (DDFS) in both arms and according to stratified subpopulations. | 5 years
  DDFS is defined as the time period between registration and first event and will be analyzed after the end of the study by referring to data from GBG patient's registry.
Invasive disease-free survival (IDFS) in both arms and according to stratified subpopulations. | 5 years
  IDFS is defined as the time period between registration and first event and will be analyzed after the end of the study by referring to data from GBG patient's registry.
Overall survival (OS) in both arms and according to stratified subpopulations. | 5 years
  OS is defined as the time period between registration and first event and will be analyzed after the end of the study by referring to data from GBG patient's registry.
Surgical substudy in patients with high probability for pCR | Baseline, after 4 cycles and before surgery (time frame + 3 weeks)
  If it can be shown at an interim analysis that the positive predictive value for a pCR of a negative (>=3) core biopsies before surgery in patients with complete clinical response is >90%, these patients might opt for having no further breast surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Untch, Prof MD, Principal Investigator — AGO, ASCO, DKG
Locations (1):
- Helios-Klinikum Berlin-Buch, Berlin, Germany

REFERENCES:
- [Background] Loibl S, von Minckwitz G, Schneeweiss A, Paepke S, Lehmann A, Rezai M, Zahm DM, Sinn P, Khandan F, Eidtmann H, Dohnal K, Heinrichs C, Huober J, Pfitzner B, Fasching PA, Andre F, Lindner JL, Sotiriou C, Dykgers A, Guo S, Gade S, Nekljudova V, Loi S, Untch M, Denkert C. PIK3CA mutations are associated with lower rates of pathologic complete response to anti-human epidermal growth factor receptor 2 (her2) therapy in primary HER2-overexpressing breast cancer. J Clin Oncol. 2014 Oct 10;32(29):3212-20. doi: 10.1200/JCO.2014.55.7876. Epub 2014 Sep 8. PMID 25199759
- [Background] Huober J, von Minckwitz G, Denkert C, Tesch H, Weiss E, Zahm DM, Belau A, Khandan F, Hauschild M, Thomssen C, Hogel B, Darb-Esfahani S, Mehta K, Loibl S. Effect of neoadjuvant anthracycline-taxane-based chemotherapy in different biological breast cancer phenotypes: overall results from the GeparTrio study. Breast Cancer Res Treat. 2010 Nov;124(1):133-40. doi: 10.1007/s10549-010-1103-9. Epub 2010 Aug 10. PMID 20697801
- [Background] Gradishar WJ, Krasnojon D, Cheporov S, Makhson AN, Manikhas GM, Clawson A, Bhar P. Significantly longer progression-free survival with nab-paclitaxel compared with docetaxel as first-line therapy for metastatic breast cancer. J Clin Oncol. 2009 Aug 1;27(22):3611-9. doi: 10.1200/JCO.2008.18.5397. Epub 2009 May 26. PMID 19470941
- [Result] Untch M, Jackisch C, Schneeweiss A, Conrad B, Aktas B, Denkert C, Eidtmann H, Wiebringhaus H, Kummel S, Hilfrich J, Warm M, Paepke S, Just M, Hanusch C, Hackmann J, Blohmer JU, Clemens M, Darb-Esfahani S, Schmitt WD, Dan Costa S, Gerber B, Engels K, Nekljudova V, Loibl S, von Minckwitz G; German Breast Group (GBG); Arbeitsgemeinschaft Gynakologische Onkologie-Breast (AGO-B) Investigators. Nab-paclitaxel versus solvent-based paclitaxel in neoadjuvant chemotherapy for early breast cancer (GeparSepto-GBG 69): a randomised, phase 3 trial. Lancet Oncol. 2016 Mar;17(3):345-356. doi: 10.1016/S1470-2045(15)00542-2. Epub 2016 Feb 8. PMID 26869049
- [Derived] Fasching PA, Szeto C, Denkert C, Benz S, Weber K, Spilman P, Budczies J, Schneeweiss A, Stickeler E, Schmatloch S, Jackisch C, Karn T, Sinn HP, Warm M, van Mackelenbergh M, Rabizadeh S, Schem C, Heinmoller E, Mueller V, Marme F, Soon-Shiong P, Nekljudova V, Untch M, Loibl S. Inferred Immune-Cell Activity Is an Independent Predictor of HER2-Negative Breast Cancer Prognosis and Response to Paclitaxel-Based Therapy in the GeparSepto Trial. Clin Cancer Res. 2023 Jul 5;29(13):2456-2465. doi: 10.1158/1078-0432.CCR-22-2213. PMID 37014668
- [Derived] Denkert C, Seither F, Schneeweiss A, Link T, Blohmer JU, Just M, Wimberger P, Forberger A, Tesch H, Jackisch C, Schmatloch S, Reinisch M, Solomayer EF, Schmitt WD, Hanusch C, Fasching PA, Lubbe K, Solbach C, Huober J, Rhiem K, Marme F, Reimer T, Schmidt M, Sinn BV, Janni W, Stickeler E, Michel L, Stotzer O, Hahnen E, Furlanetto J, Seiler S, Nekljudova V, Untch M, Loibl S. Clinical and molecular characteristics of HER2-low-positive breast cancer: pooled analysis of individual patient data from four prospective, neoadjuvant clinical trials. Lancet Oncol. 2021 Aug;22(8):1151-1161. doi: 10.1016/S1470-2045(21)00301-6. Epub 2021 Jul 9. PMID 34252375
- [Derived] Furlanetto J, Jackisch C, Untch M, Schneeweiss A, Schmatloch S, Aktas B, Denkert C, Wiebringhaus H, Kummel S, Warm M, Paepke S, Just M, Hanusch C, Hackmann J, Blohmer JU, Clemens M, Costa SD, Gerber B, Nekljudova V, Loibl S, von Minckwitz G. Efficacy and safety of nab-paclitaxel 125 mg/m2 and nab-paclitaxel 150 mg/m2 compared to paclitaxel in early high-risk breast cancer. Results from the neoadjuvant randomized GeparSepto study (GBG 69). Breast Cancer Res Treat. 2017 Jun;163(3):495-506. doi: 10.1007/s10549-017-4200-1. Epub 2017 Mar 17. PMID 28315068
- See also: Sponsor study homepage — https://www.gbg.de/de/studien/